CLINICAL TRIAL: NCT04549376
Title: Virucidal Effect of Povidone Iodine on COVID-19 In-Vivo: an Open Label Randomized Clinical Trial
Brief Title: Virucidal Effect of Povidone Iodine on COVID-19 In-Vivo
Acronym: VEP-COV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DR. MALA KHAN (Other Government)
Collaborators: Dhaka Medical College (Other)
Responsible Party: Sponsor-Investigator, DR. MALA KHAN, Director General, Bangladesh Reference Institute of Chemical Measurements (BRICM)
Organization: Bangladesh Reference Institute of Chemical Measurements (BRICM) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BRiCM-1131-2020
Record Dates: First submitted 2020-09-11; First posted 2020-09-16 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: COVID19
Keywords: COVID19; prevention; Povidone Iodine; Low and middle income countries
MeSH Terms: conditions — COVID-19 | interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- PVP-I 0.4% NI (Experimental): Arm-1 will receive Povidone iodine (PVP-I) nasal irrigation (NI) at concentration of 0.4% single time
  Interventions: Drug: Povidone-Iodine 0.4% NI
- PVP-I 0.5% NI (Experimental): Arm-2 will receive Povidone iodine (PVP-I) nasal irrigation at concentration of 0.5% single time
  Interventions: Drug: Povidone-Iodine 0.5% NI
- PVP-I 0.6% NI (Experimental): Arm-3 will receive Povidone iodine (PVP-I) nasal irrigation at concentration of 0.6% single time
  Interventions: Drug: Povidone-Iodine 0.6% NI
- PVP-I NS 0.5% NS (Experimental): Arm-4 will receive will receive PVP-I nasal spray (NS) at concentration of 0.5% single time
  Interventions: Drug: Povidone-Iodine 0.5% NS
- PVP-I 0.6% NS (Experimental): Arm-5 will receive will receive PVP-I nasal spray at concentration of 0.6% single time
  Interventions: Drug: Povidone-Iodine 0.6% NS
- DW NI (Placebo Comparator): Arm-6 will receive distilled water through nasal irrigation
  Interventions: Other: Placebo comparator: DW-NI
- DW NS (Placebo Comparator): Arm-7 will receive distilled water through nasal spray
  Interventions: Other: Placebo comparator: DW-NS

INTERVENTIONS:
Drug: Povidone-Iodine 0.4% NI — Povidone iodine (PVP-I) nasal irrigation at concentration of 0.4%
  Other Names: Povidone-Iodine 0.4%
  Arms: PVP-I 0.4% NI
Drug: Povidone-Iodine 0.5% NI — Povidone iodine (PVP-I) nasal irrigation at concentration of 0.5%
  Other Names: Povidone-Iodine 0.5%
  Arms: PVP-I 0.5% NI
Drug: Povidone-Iodine 0.6% NI — Povidone iodine (PVP-I) nasal irrigation at concentration of 0.6%
  Other Names: Povidone-Iodine 0.6%
  Arms: PVP-I 0.6% NI
Drug: Povidone-Iodine 0.5% NS — Povidone iodine (PVP-I) nasal spray at concentration of 0.5%
  Other Names: Povidone-Iodine 0.5%
  Arms: PVP-I NS 0.5% NS
Drug: Povidone-Iodine 0.6% NS — Povidone iodine (PVP-I) nasal spray at concentration of 0.6%
  Other Names: Povidone-Iodine 0.6%
  Arms: PVP-I 0.6% NS
Other: Placebo comparator: DW-NI — Nasal irrigation will be provided by Distilled water
  Other Names: Distilled water (DI) in the form of Nasal Irrigation
  Arms: DW NI
Other: Placebo comparator: DW-NS — Nasal spray will be provided by Distilled water
  Other Names: Distilled water (DI) in the form of Nasal spray
  Arms: DW NS

SUMMARY:
It is an established fact that, corona virus spread through the respiratory droplets. Colonization of the virus in oropharynx and/or nasopharynx is considered to be major factor for transmissibility of the virus through respiratory secretions. Preventing colonization of the virus by administrating povidone iodine in the nasal passage therefore, a rational thought which is supported by recent evidence of in-vitro virucidal action of povidone iodine in Severe Acute Respiratory Syndrome-Coronavirus 2 (SARS CoV-2). Therefore, the study is designed to assess the virucidal effect of povidone iodine on COVID-19 virus in-vivo.This open label randomized clinical trial will be conducted at Department of Otorhinolaryngology and Head Neck Surgery, in collaboration with Department of Virology and Department of Medicine in Dhaka Medical College (DMC) Hospital. The study will be conducted from September 2020 to October 2020. Total 175 confirmed cases of COVID-19 disease, proven by Reverse transcription polymerase chain reaction (RT-PCR) testing will be enrolled in this study. Written informed consent will be ensured before participation. In case of no literacy, finger print will be considered for written permission.Consent will be sought from the legal guardian in case of minor or underaged.Formal ethical clearance will be taken from Ethical Review Committee (ERC) of Dhaka Medical College. All of the Participants will be divided into seven groups: Group A will receive Povidone iodine (PVP-I) nasal irrigation at concentration of 0.4%, Group B and Group C will received 0.5% and 0.6%; Group D will receive PVP-I nasal spray at concentration of 0.5% and Group E will received at 0.6% concentration. Group F (Placebo comparator group) will receive nasal irrigation by distilled water (DW) and Group G (Placebo comparator group) will received nasal spray by distilled water. The contact time will be minimum 30 seconds. After the individual application of PVP-I and distilled water in respective participant, they will be tested again for RT-PCR for COVID-19 from nasopharyngeal and oropharyngeal sample. All patients will be subjected to detail history, physical examination and adverse events. Block Randomization will be followed for randomization. Data will be recorded in a semi-structured questionnaire and will be analyzed by 'R-4.0.2' data analysis software

DETAILED DESCRIPTION:
Rationale of the study

The coronavirus disease 2019 (COVID-19) is a highly infectious disease and cause human to human transmission primarily by respiratory droplets from coughing, sneezing and speaking. In early SARS-CoV-2 infection, a greater viral titre can be found in saliva and nasal mucous; minimization of these titres should help to reduce cross infection. Povidone-iodine (PVP-I) disinfectant has better anti-viral activity than other antiseptics and has already been proven to be an extremely effective virucide in vitro against severe acute respiratory syndrome and Middle East respiratory syndrome coronaviruses (SARS-CoV and MERS-CoV). Its' in vivo virucidal activity is unknown, though its nasal or oral preparation can be effective in reducing transmission. Earlier, a very few studies have evaluated the efficacy of povidone-iodine as nasal antiseptics or oral rinse antiseptics against the SARS-CoV-2 virus but the result of those studies are not undebatable. So aim of this study is to investigate the virucidal activity of povidone iodine on coronavirus located on the mucosal surface of oropharynx and nasopharynx and is very rational in this pandemic period.

Research Hypothesis:

Objectives:

General Objective:

To determine the virucidal efficacy of povidone iodine on COVID-19 virus located in nasopharynx.

Secondary objectives:

i. To determine the efficacy of povidone iodine to clear COVID-19 virus located in nasopharynx ii. To assess the adverse events among the groups

Study Design: Open label randomized clinical trial. Place of Study: Department of Otorhinolaryngology and Head Neck Surgery, in collaboration with Department of Virology and Department of Medicine, Dhaka Medical College Hospital, Dhaka, Bangladesh.

Period of study: The study period will be September 2020 to November 2020. Study population: Confirmed cases of COVID-19 disease proven by RT-PCR testing. Sampling and Statistical basis of the sample size: The sample size is determined using the following formula Sample size: estimated sample size 189 (twenty seven in each group) Research instruments General questionnaire for recording baseline information A checklist for for detecting COVID-19 status

Method and data collection:

Participant selection and enrollment: All patients admitted to the medical wards through emergency department or Outpatient department with suspected COVID-19 cases will be initially approached and screened for confirmation of the COVID-19. Confirmation of the COVID-19 will be done by positive impression of RT-PCR result. Following confirmation of the viral infection, the patients will be seen by the ward doctors and clinical trial physicians (registered physicians). Moreover, baseline complete blood count (CBC) will be done for each patient. Chest X-ray/High resolution computed tomography (HRCT) will be done in necessary case. The ward doctors and trial physicians will together care for the patient; then the patients will be briefed about the aim, objective and details of the procedure of the study. If without capacity, their relatives will be approached about the trial and seek their consent for recruitment. As this study will be confined into a tertiary care hospital, patients will be recruited up to day 4 of illness.

Consenting participants: It will be prioritized that the patients will be treated early for COVID-19 management by standard regiment and in accordance to the guidance of the national guidelines. And within shortest possible time preferably within 4 hours of admission, consenting procedure will be completed either from the patient or from the attendant/legal guardian of the patients to obtain the full potential benefit of the treatment. Written informed consent will be obtained from the patient in their own language [Bengali] by trial physicians working on the trial.

Screening for eligibility: During admission, demographic and clinical details including name, age/date of birth, gender, duration of onset of fever and hospitalization, vital statistics will be recorded before randomization. RT PCR for COVID-19 will be used for confirmation of the COVID-19 virus infection. A screening log will be maintained including these essential details and the decision taken by the patient or attendant or legal guardian where appropriate concerning recruitment. Ineligible and non-recruited patients will also be cared by the ward physicians following standard treatment guidelines.

Procedure of randomization: The study participants will be randomly assigned in this study into six equal groups; where each group has equal opportunity to receive any treatment option. Randomization will be done by block randomization methods. Randomization will be done quickly, with baseline information typically captured in <15 min. Recruitment & randomization will be performed contemporaneously with assessment/resuscitation of patients by a second person so that medical care is not delayed by recruitment. Patients will only be randomized once baseline data has been entered; after this has been done, participants will not be withdrawn from the study. Following completion of the randomization, the trial physicians reported the Principal Investigator (PI) of the trial and then the Principal Investigator (PI) handed over an opaque sealed envelope, which will be numbered sequentially to correspond to patient enrollment numbers, which will be used for concealment of treatment allocations. Envelopes will be kept in a locked drawer and will be opened in strictly numerical order by in supervisor in presence of nursing supervisor of study unit. Allocation between arms will initially be equal, although this may be revised following guidance of the PI and his team (as per the statistical plan).

Withdrawal of study participants: Participants are free to withdraw from the study at any point, for any reason. If this occurs, the primary reason for withdrawal will be documented in the participant's case record form. The participant will have the option of withdrawal from:

participant samples. Randomized patients who wish to withdraw from the study before they have undertaken any study-related procedures will be replaced. Data on the original participant will be kept on the CRF/database if the participant agrees to this.

Investigational medicinal products:

All of the Participants will be divided into three groups: Group A will receive Povidone iodine (PVP-I) nasal irrigation (NI) at three different concentration of 0.4%, Group B and Group C will received 0.5% and 0.6%; Group D will receive PVP-I nasal spray (NS) at concentration of 0.5% and Group E will received at 0.6% concentration. Group F (Placebo comparator group) will receive nasal irrigation by distilled water and Group G (Placebo comparator group) will received nasal spray by distilled water Participant compliance: The study team will not create any problem with compliance while the patient is under care and supervision in hospital. It was ensured that all recruited patients receive the appropriate interventions, although it could be interrupted due to the onset of potential adverse effects such as hypotension.

Responsibility sharing of care of the patients: As the patients will remain under the care of the hospitals' consultant physicians/unit head who will have primary responsibility for their management. Management protocols will be agreed between the medical team and study team. Decisions about intubation, requirement of blood and blood products, transfer of patients to intensive care, weaning of ventilation and extubation will be made by the medical team independently of study doctors. All decisions will be based on the patient's clinical condition and the available hospital resources, as per usual hospital practice. The study team preferably by trial physicians will note down the record in patient's Case Record Form (CRF).

Methods of data collection: data collection will be done by the trial physicians. A paper based semi-structured questionnaire was made and pre-tested before data collection. All potential participants will be recorded in this database at first contact and assigned a study number. This study number (eg DMC-PVP-I-0001) will be used for all data and samples collected from that person. Study doctors will recruit and randomize patients at the bedside with a randomization procedure. They will not be able to predict allocation before randomization. Following randomization, allocation will be done by the PI and trial physicians or nurse will confirm the administration of the either drug/distilled water. Patients will be closely monitored. Temperature will be measured in every 6 hours, blood pressure, respiratory rate, pulse rate will be measured in every hour. Urine output will be measured in every 8 hours. Drug related side effects or any adverse events will be observed in each group.

If there is no reaction or unusual event, another RT-PCR sample will be collected from the nasopharynx and sent for further testing.

Total duration of the follow up will be for 2 days (or person fulfills the discharge criteria). All clinical events will be noted in case record form by trial physicians, including vital status at hospital discharge. Data entry will be date/time stamped. Laboratory analysis data will be collected using same CRF.

Data quality and standards: following collection, all data set and collected record form will be checked. A formal clinical data management plan will be written before the study starts, agreed by the co-investigators, and Data Monitoring Committee, and documented trail master file. Laboratory results will be discussed regularly between the PI and laboratory managers.

Proposed Analysis Plan of the study:

Data analysis will be done by data management software, R-4.0.2'. Statistical significance is set as 95% confidence level at 5% acceptable error level. Differences will be considered significant at the P < 0.05 level for all these tests. The data will be expressed as means ±Standard deviations (SD) for continuous variables and as frequencies (%) for categorical variables. Chi-square test, student t test or ANOVA or other statistical test will be used in case of normally distributed data and similar non-parametric data will be used whenever appropriate. Graph & chart will be expressed by Microsoft Excel 2016.

Ethical consideration:

The researcher is duly concern about the ethical issues relate to the study. In this study the following criteria will be followed to ensure maintaining the ethical values. All ethical measure will be followed in accordance to the current Declaration of the Helsinki and Good clinical practice (GCP) and Good laboratory practice (GLP) guidelines.

Facilities available at study center:

The RT-PCR and other study-related testing will be done at DMCH. DMCH was designated as a COVID dedicated hospital which provide multidisciplinary care.Necessary investigations are available here with minimal cost.

ELIGIBILITY:
Inclusion Criteria:

* Age: 15-90 years
* Either gender
* Patients diagnosed with COVID-19 disease by RT-PCR
* Have confirmed COVID-19 symptoms and symptom onset within the past 10 days
* Capable of using a nasal spray device and perform nasal irrigation required by the study
* Willing to participate

Exclusion Criteria:

* Patient with known sensitivity to PVP-I aqueous antiseptic solution or any of its listed excipients
* Previously diagnosed thyroid disease
* Patients with chronic renal failure (stage ≥3 by estimated Glomerular Filtration rate (eGFR) Modification of Diet in Renal Disease( MDRD)
* Patients with acute renal failure (KDIGO ≥stage 2: creatinine ≥2 X baseline)
* Pregnant and lactating mother
* Current requirement for invasive or non-invasive ventilation or planned within next 6 hours.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Proportion of COVID-19 positive cases following intervention | 5 minutes-30 minutes
  Proportion of COVID-19 positive cases following intervention in all groups

SECONDARY OUTCOMES:
Adverse events | 1 minute to 24 hours
  Any adverse event following administration of both intervention and placebo agent

CONTACTS AND LOCATIONS:
Overall Officials: Prof Sk Nurul Fattah Rumi, MBBS, MS, Study Chair — Dhaka Medical College
Locations (1):
- Dhaka Medical College, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
After completion of the project, a manuscript will be prepared and will be shared to the journal authority for publication. Data will be shared with the journal authority and make public as part of the publication.
Supporting Information: SAP, ICF, CSR
Time Frame: 6 months
Access Criteria: Available on public domain like figshare, researchgate and others

REFERENCES:
- [Derived] Kamal Arefin M, Banu SS, Nasir Uddin AKM, Nurul Fattah Rumi SK, Khan M, Kaiser A, Arafat MS, Chowdhury JA, Khan MAS, Hasan MJ. Virucidal Effect of Povidone Iodine on SARS-CoV-2 in Nasopharynx: An Open-label Randomized Clinical Trial. Indian J Otolaryngol Head Neck Surg. 2022 Oct;74(Suppl 2):3283-3292. doi: 10.1007/s12070-022-03106-0. Epub 2022 May 6. PMID 35572740
- [Derived] Hasan MJ, Rumi SKNF, Banu SS, Uddin AKMN, Islam MS, Arefin MK. Virucidal effect of povidone iodine on COVID-19 in the nasopharynx: A structured summary of a study protocol for an open-label randomized clinical trial. Trials. 2021 Jan 4;22(1):2. doi: 10.1186/s13063-020-04963-2. PMID 33397432